CLINICAL TRIAL: NCT02187432
Title: The Eurocyst Initiative: Building a Reference Center Network Across EUROpe to Establish a Large-scale Longitudinal Observational Cohort of Autosomal Dominant polyCYSTic Kidney Disease (ADPKD) Patients
Brief Title: The Eurocyst Initiative: Building a Network of ADPKD Reference Centers Across Europe
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Andreas L. Serra (Other)
Responsible Party: Sponsor-Investigator, Andreas L. Serra, MD, University of Zurich
Organization: University of Zurich (Other)
Other Study IDs: Eurocyst
Record Dates: First submitted 2014-02-24; First posted 2014-07-11 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The following samples will be collected: blood, spot urine and 24h urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ADPKD: EuroCYST is and observational trail aiming to investigate disease progression across the different stages of disease and stage specific morbidity and mortality factors in a longitudinal observational multi center study and to evaluate the levels of and associations between the impacts of patients reported disease outcome (quality of life (QoL), pain, self-estimated health status, health burden).

SUMMARY:
EuroCYST initiative aims to build a large, well-characterized cohort of Autosomal Dominant polyCYSTic Kidney Disease (ADPKD) subjects who are followed in a longitudinal observational cohort study has the potential to identify progression factors and biomarkers, and to assess disease stage specific mortality, morbidity and health care costs.

DETAILED DESCRIPTION:
The EuroCYST Initiative aims to build a network of ADPKD reference centers across Europe and to establish a large-scale observational cohort of ADPKD patients for the purpose of studying the pathogenesis, rate of disease progression, progression rate modifiers, disease stage specific morbidity, mortality, health economic issues and the predictive value of biomarkers in ADPKD. Overall 1,100 patients will be enrolled in 14 study sites across Europe and will be followed up for at least three years. The ADPKD reference center network across Europe and the observational cohort study will enable European ADPKD researchers to gain insight into the natural history, heterogeneity and associated complications of the disease as well as how it affects the lives of patients across Europe.

ELIGIBILITY:
Inclusion Criteria:

* Participants ≥ 18 years;
* Clinical diagnosis of ADPKD based on kidney imaging and family history;
* Estimated Glomerular Filtration Rate (eGFR) ≥ 30 ml/min/1.73m2 (Chronic Kidney Disease Epidemiology Collaboration(CKD-EPI)- formula);
* Provided written informed consent.

Exclusion Criteria:

* Receiving chronic renal replacement therapy before enrollment (dialysis, allograft) or anticipated in the following 12 months after enrollment;
* Participation in a clinical trial aiming to modify disease outcome one year or less before enrollment in the EuroCYST study;
* New York Heart Association (NYHA) stadium IV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include 1,100 participants aged 18 and above with a diagnosis of ADPKD, diagnosed via imaging and family history. The assessment of participants is based on defined inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2013-08; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
disease progression | participants will be followed annually for at least 3 years
  Investigate disease progression and association of disease biomarkers with the onset and severity of ADPKD-related outcomes.

SECONDARY OUTCOMES:
QOL (Quality of Life) | participants will be followed annually for at least 3 years
  Evaluate and establish the level of disease impact on self-estimated health status, pain, QoL, socioeconomic status (SES), ADPKD-related health burden, health care resource use.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas L Serra, MD, Principal Investigator — University of Zurich
Locations (14):
- Cliniques universitaires Saint-Luc, Brussels, Belgium
- Charles University Prague, Prague, Czechia
- France (2):
  - Centre hospitalier universitaire de Brest, Brest
  - Hôpital de Rangueil, Toulouse
- Germany (3):
  - Charité Universitätsmedizin Berlin, Berlin
  - University Hospital Erlangen, Erlangen
  - University Hospital Freiburg, Freiburg im Breisgau
- Istituto di Ricerche Farmacologiche "Mario Negri", Bergamo, Italy
- University Medical Center Groningen, Groningen, Netherlands
- Fundació Puigvert, Barcelona, Spain
- University Hospital Zurich, Zurich, Switzerland
- Istanbul School of Medicine, Istanbul, Turkey (Türkiye)
- United Kingdom (2):
  - University of Cambridge, Cambridge Cancer Center, Cambridge
  - University of Sheffield Medical School Academic Unit of Nephrology Department of Infection and Immunity, Sheffield